CLINICAL TRIAL: NCT06597435
Title: Effect of Product Characteristics on the Appeal and Sensory Attributes of Nicotine Pouches
Brief Title: Effects of Nicotine Pouch Characteristics on Perceptions and Behavior
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Dae Hee Han, Postdoctoral Fellow, University of Southern California
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: UP-23-01161; K99DA058241 (NIH)
Record Dates: First submitted 2024-08-29; First posted 2024-09-19 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-09

CONDITIONS: Nicotine Pouch Self-Administration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Nicotine pouch containing high nicotine (6-8mg) (Experimental): Participants will self-administer a nicotine pouch containing 6-8mg nicotine.
  Interventions: Other: Nicotine pouch
- Nicotine pouch containing low nicotine (3-4mg) (Placebo Comparator): Participants will self-administer a nicotine pouch containing 3-4mg nicotine.
  Interventions: Other: Nicotine pouch
- Nicotine pouch with low pH (less than 8.5) (Experimental): Participants will self-administer a nicotine pouch with low pH (less than 8.5).
  Interventions: Other: Nicotine pouch
- Nicotine pouch with high pH (8.5 or greater) (Placebo Comparator): Participants will self-administer a nicotine pouch with high pH (8.5 or greater).
  Interventions: Other: Nicotine pouch

INTERVENTIONS:
Other: Nicotine pouch — Participants will self-administer an experimenter-provided nicotine pouch

SUMMARY:
There is a growing sector of modern tobacco-free oral nicotine pouches that are federally regulated as non-medicinal nicotine/tobacco products. While nicotine pouches employ marketing approaches that may attract current tobacco users, such as marketing themes connoting minimal harm, information on the long-term health effects of nicotine pouches is lacking. nicotine pouches may appeal to younger adults because they are available in similar product characteristics (e.g., nicotine concentration, protonated nicotine) that many younger people prefer to use in e-cigarettes. In addition, nicotine pouches may be of particular interest to younger adult e-cigarette users because these products can be used discreetly where vaping is not allowed, which may translate into an increased likelihood of becoming dual users of e-cigarettes and nicotine pouches. Indeed, approximately 15% young adults who used e-cigarettes in the past 30 days were past 30-day nicotine pouch users. Manufacturers of modern nicotine pouches use acid additives to lower pH, which changes nicotine from a free-base to a protonated nicotine, resulting in improved appeal and sensory experience and higher abuse liability. Thus, nicotine concentration and pH in modern nicotine pouches should be focal targets for regulatory policies. Evidence is also lacking on mechanisms mediating differences in product appeal and abuse liability of nicotine pouches across products varying in nicotine concentration and pH level. The scientific objective of this research is to assess the effect of variation in nicotine concentration in nicotine pouches and its interaction effect with pH level on the proximal outcomes of relevance to the U.S. Food and Drug Administration regulation: sensory attributes and product appeal among younger adults who use nicotine pouches in the past 30 days (current dual users of nicotine pouches and e-cigarettes and/or combustible cigarettes will be eligible) and are unmotivated to quit nicotine use. This innovative project proposes to conduct a double-blind within-subject randomized study in which participants (N = 72) will administer nicotine pouches varied by nicotine concentration (e.g., 3 vs 6 mg) and pH (e.g., 8.5 or greater vs. less than 8.5) to achieve the project aim: to evaluate the effects of nicotine concentration and pH on subjective product appeal and sensory attributes of nicotine pouches. The findings of this proposed research will provide the U.S. Food and Drug Administration with new evidence necessary to inform regulatory restrictions on product characteristics and constituents of nicotine pouches, which may put young adults at risk of using a novel class of oral nicotine products.

DETAILED DESCRIPTION:
The project will assess the effect of variation in nicotine concentration in nicotine pouches and its interaction effect with pH level on two proximal outcomes of relevance to regulation: (1) sensory attributes and (2) product appeal in an experimental study of young adult (21-35 years) nicotine pouch users who are unmotivated to quit nicotine use. Before the experimental session, the investigators will conduct orientation sessions where participants will confirm age, provide informed consent, and complete verification of nicotine use status by cotinine test strip. Eligible participants will be scheduled for their experimental visits and instructed to abstain from nicotine use for 8 hours (overnight) prior to the experimental session. During the experimental session, participants (N=72) will self-administer 4 different nicotine pouches varied by nicotine concentration (e.g., 3mg vs. 6mg) and pH (e.g., 8.5 or greater vs. less than 8.5) equated on other product characteristics (e.g., pouch size and weight, moisture content) in a single-visit 4-hour within-subject double-blind randomized clinical trial. Participants will rate the appeal (e.g., liking, disliking, willingness to use again) and sensory attributes (e.g., smoothness, harshness, sweetness, bitterness, irritation) of each nicotine pouch and select their favorite nicotine pouch product (alternative appeal measure) at the end of the study. During the experimental sessions, questionnaires will also assess participants' nicotine product use characteristics and sociodemographic characteristics. After the experimental session, participants will be remunerated. Study materials will be selected among commercially available products manufactured by leading providers (e.g., ZYN, Lucy, VELO, Rogue, on!), and product constituents will be analyzed and reported. This project will identify two product characteristics (low pH and high nicotine) that may perpetuate nicotine pouch use and nicotine dependence risk by increasing their appeal and potential abuse liability in young adults, and therefore merit targeting in the U.S. Food and Drug Administration regulation.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 21-35 years old.
* Current nicotine pouch users (used nicotine pouches in the past 30 days). Current dual users of nicotine pouches and e-cigarettes and/or combustible cigarettes will be eligible.
* Positive cotinine test via saliva test strip.
* Unmotivated to quit nicotine use.
* English language competency (read and speak English). The instruments used have not been translated and/or validated for other languages.

Exclusion Criteria:

* Intention to quit nicotine use in the next 30 days.
* Current pregnancy or breastfeeding (urine pregnancy test will be conducted during the orientation session).
* History of stroke, seizures, high blood pressure (hypertension), heart disease/problems, lung disease/lung problems, or cardiovascular disease contraindications for nicotine.
* People under 21 years will be excluded to correspond with the legal age for purchasing tobacco products in the United States. Special subject populations will not be recruited.

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Subjective Appeal and sensory experience | During the 3-hour experimental session, participant will self-administer 4 nicotine pouches, each with a 5-minute administration period. There will a 40-minute inter-product rest interval.
  Self-report measures of product appeal (e.g., liking, disliking, willingness to use again) and sensory attributes (e.g., sweetness, smoothness, bitterness, harshness) will be completed following the nicotine pouch administration.

CONTACTS AND LOCATIONS:
Overall Officials: Dae Hee Han, PhD, Principal Investigator — University of Southern California
Locations (2):
- United States (2):
  - University of Southern California, Los Angeles, California
  - University of Southern California - Clinical Sciences Building, Los Angeles, California